CLINICAL TRIAL: NCT07000032
Title: A Longitudinal Study on Dysphagia and Associated Nutritional Complications Following Oral Cancer Surgery
Brief Title: The Swallowing Function of Oral Cancer Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending anesthesiologist, National Taiwan University Hospital
Other Study IDs: 202501062RINA
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: The Swallowing Changes
Keywords: oral cancer surgery; swallowing; nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For investigating the specific nutrition gene
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing oral cancer surgery: patients undergoing oral cancer surgery
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — This is an observational cohort

SUMMARY:
This study enrolled patients who underwent oral cancer resection. Swallowing function, muscle status, and nutritional status were assessed before treatment, one month after treatment, and between three months to one year post-treatment.

DETAILED DESCRIPTION:
Dysphagia is a common and debilitating symptom among patients who undergo oral cancer resection with reconstruction followed by adjuvant radiotherapy. During the course of the disease, approximately 20% to 98% of patients experience swallowing difficulties. This is primarily caused by tumor destruction, postoperative sequelae from surgical resection, and the adverse effects of radiotherapy and chemotherapy. The use of chemotherapy or radiotherapy-particularly when combined-increases the incidence of complications such as oropharyngeal mucositis, odynophagia, dysgeusia, xerostomia, nausea, vomiting, and fatigue. These complications may lead to dehydration and significant weight loss, which in turn negatively impact nutritional status, functional ability, and quality of life.

This study enrolled patients who underwent oral cancer surgery. Swallowing function, muscle status, and nutritional status were assessed before treatment, one month after treatment, and between three months to one year post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing oral cancer

Exclusion Criteria:

* patients unable to unable to cooperate with the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing oral cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
bolus presence time | one year after surgery
  The opening of hypopharynx

IPD SHARING:
Plan to Share IPD: No
Due to ethical issue